CLINICAL TRIAL: NCT00156650
Title: Male Hormonal Contraception Development: Suppression of Spermatogenesis With the Addition of a Potent GnRH Antagonist (Acyline) to Testosterone and DMPA (ACY-5) -Sub-Study (HOP 5)
Brief Title: Manipulation of the Intratesticular Hormonal Milieu With Exogenous Testosterone (HOP 5) Testicular Aspiration Addendum
Acronym: IHOP-5
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: William J Bremner, MD, PhD, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 04-0832-D-substudy; U54HD042454 (NIH)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Contraception
Keywords: Male contraception; Testosterone
MeSH Terms: interventions — acyline; Testosterone; Medroxyprogesterone Acetate; N,N-dimethyl-4-anisidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Testosterone (T) gel for 6 months + DMPA (Depo-Medroxyprogesterone) (injected into muscle Day 0 & at Month 3)
  Interventions: Drug: Testosterone Gel; Drug: Depo-Medroxyprogesterone
- 2 (Active Comparator): T gel for 6 months + DMPA (Day 0 & Month 3) + Acyline 300 mcg/kg twice monthly for 12 weeks
  Interventions: Drug: Acyline; Drug: Testosterone Gel; Drug: Depo-Medroxyprogesterone

INTERVENTIONS:
Drug: Acyline — Acyline 300 mcg/kg SQ(Subcutaneously)twice monthly for 12 weeks
  Arms: 2
Drug: Testosterone Gel — Testosterone (T) gel 10 g daily for 6 months
  Other Names: Testim
Drug: Depo-Medroxyprogesterone — 300 mg IM every 3 months
  Other Names: DMPA

SUMMARY:
This study is being offered to all participants of the ACY-5 study as an optional addition to the male contraceptive study in which they participated. Participation is voluntary.

The purpose of this added procedure (Testicular Aspiration-HOP 3) is to determine the amount of testosterone (male hormone) in the testes of men who are on a male contraceptive regimen.

DETAILED DESCRIPTION:
The goal of our contraception study (ACY-5) is to develop a hormonal regimen where in all individuals enrolled achieve azoospermia (zero sperm). However, early data demonstrated that some individuals have persistent sperm in their semen despite treatment. We hope to be able to determine whether differences in intratesticular hormone levels account for persistent sperm production in men who do not reach counts of zero as compared to those who do in the male contraceptive study. This study will measure testosterone levels in the testes of men who are participating in male contraceptive studies. Testosterone will be measured in a small amount of testicular fluid at the end of the study treatment phase after sperm counts have been reduced to zero or very low levels.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18-55
* In good health
* With normal sperm counts and willing to use an acceptable form of contraception during the study

Exclusion Criteria:

* Male in poor health
* Significant chronic or acute medical illness
* Skin conditions that might interfere with or be exacerbated by testosterone gel
* No history of alcohol, illicit drug or anabolic steroid abuse
* Abnormal reproductive function
* Participation in a long-term male contraceptive study within three months of screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2004-12; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Intratesticular hormone levels | One year

SECONDARY OUTCOMES:
sperm count levels | One year

CONTACTS AND LOCATIONS:
Overall Officials: William Bremner, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Coviello AD, Bremner WJ, Matsumoto AM, Herbst KL, Amory JK, Anawalt BD, Yan X, Brown TR, Wright WW, Zirkin BR, Jarow JP. Intratesticular testosterone concentrations comparable with serum levels are not sufficient to maintain normal sperm production in men receiving a hormonal contraceptive regimen. J Androl. 2004 Nov-Dec;25(6):931-8. doi: 10.1002/j.1939-4640.2004.tb03164.x. PMID 15477366
- [Background] Coviello AD, Matsumoto AM, Bremner WJ, Herbst KL, Amory JK, Anawalt BD, Sutton PR, Wright WW, Brown TR, Yan X, Zirkin BR, Jarow JP. Low-dose human chorionic gonadotropin maintains intratesticular testosterone in normal men with testosterone-induced gonadotropin suppression. J Clin Endocrinol Metab. 2005 May;90(5):2595-602. doi: 10.1210/jc.2004-0802. Epub 2005 Feb 15. PMID 15713727
- [Result] Page ST, Kalhorn TF, Bremner WJ, Anawalt BD, Matsumoto AM, Amory JK. Intratesticular androgens and spermatogenesis during severe gonadotropin suppression induced by male hormonal contraceptive treatment. J Androl. 2007 Sep-Oct;28(5):734-41. doi: 10.2164/jandrol.107.002790. Epub 2007 May 9. PMID 17494097